CLINICAL TRIAL: NCT07028411
Title: The Effectiveness of the Board Game on Primary Healthcare Nurses' Knowledge, Attitudes, and Confidence in Dengue-related Practice: a Cluster Randomized Controlled Trial
Brief Title: The Effectiveness of the Board Game on Primary Healthcare Nurses' Knowledge, Attitudes, and Confidence in Dengue-related Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Nuzul Sri Hertanti, RN, MS, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KE/FK/0902/EC/2025
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-06

CONDITIONS: Knowledge; Attitude; Confidence, Self
Keywords: board game; dengue; knowledge; attitude; confidence; nurse
MeSH Terms: conditions — Behavior; Dengue

STUDY DESIGN:
Intervention Model Description: Two teaching methods will be implemented: an educational board game as intervention group and lecture as control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational board game (Experimental): Participants will receive an educational board game one time for 90 minutes.
  Interventions: Behavioral: Educational board game
- Lecture group (Active Comparator): Participants will receive a lecture-based intervention one time for 90 minutes.
  Interventions: Behavioral: Lecture

INTERVENTIONS:
Behavioral: Educational board game — The educational board game will be administered once for a duration of 90 minutes, consisting of a gameplay session followed by a debriefing.
  Arms: Educational board game
Behavioral: Lecture — The lecture will be administered once for a duration of 90 minutes, consisting of video lecture followed by question and answer (QnA) session.
  Arms: Lecture group

SUMMARY:
This cluster randomized controlled trial aims to evaluate the effectiveness of an educational board game compared to a lecture-based intervention on improving knowledge, attitudes, and confidence in dengue-related practice among nurses working in primary healthcare (PHC) units. Additionally, the study will assess PHC nurses' satisfaction with the learning experience. A total of 82 participants from 14 PHC unit clusters in Yogyakarta, Indonesia will be randomly assigned to either the intervention group (educational board game) or the control group (lecture-based intervention). Each group will receive a one-time 90-minute session of assigned intervention. Outcomes related to knowledge, attitudes, and confidence will be measured at multiple time points.

DETAILED DESCRIPTION:
Considering the multiple roles of PHC nurses in dengue prevention and management, there is a need for training methods that are not only informative but also actively engaging and time-efficient. Educational board games offer a promising interactive learning strategy. However, their application among healthcare professionals, particularly nurses, remains underexplored.

The main purpose of this study is to examine whether an educational board game can improve PHC nurses' knowledge, attitudes, and confidence in dengue-related practice compared to a lecture-based intervention. In addition, the study will evaluate participants' satisfaction with the learning experience.

This two-arm parallel cluster randomized controlled trial will be conducted in Yogyakarta, Indonesia, involving 82 participants from 14 PHC unit clusters. These clusters will be randomly allocated into two groups: the intervention group (educational board game) and the control group (lecture-based intervention). Each group will receive a single 90-minute educational session.

Outcomes on knowledge, attitudes, and confidence will be assessed at multiple time points. Data will be analyzed using a linear mixed-effects model (LMM) to evaluate the interaction effects between group and time. Findings from this study may offer valuable insights for healthcare institutions and policymakers to consider integrating board games into professional training and continuing professional development (CPD) programs.

ELIGIBILITY:
Inclusion Criteria:

* Full-time employed nurses in the PHC unit
* Nurses who have experience in assessing dengue-suspected patients
* Nurses who have at least three months of work experience in the current PHC unit
* Nurses who have a smartphone for online communication
* Nurses who are familiar with WhatsApp applications

Exclusion Criteria:

* Nurses on maternity or annual leave during the data collection period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2025-08-08 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Knowledge | Baseline, immediately after intervention, and follow up at one-month post intervention.
  This study will use the Indonesian version of Dengue Knowledge Questionnaire to measure PHC nurses' knowledge of dengue. The questionnaire consists of seven items, with response options of "true," "false," or "unknown." Each correct answer will receive 1 point, while incorrect or unknown responses receive 0 points. Total scores range from 0 to 7, with higher scores reflecting a better knowledge of dengue.
Attitude | Baseline, immediately after intervention, and follow up at one-month post intervention.
  The study will use the Indonesian version of Dengue Preventive Attitudes Questionnaire to measure nurses' attitudes toward dengue prevention. It consists of seven items, each rated on a five-point Likert scale, with 1 indicating "strongly disagree" and 5 indicating "strongly agree." Total scores range from 7 to 35, with higher scores representing more favorable attitudes toward dengue prevention.
Confidence | Baseline, immediately after intervention, and follow up at one-month post intervention.
  The study will use the Indonesian version of the five-item Confidence-Scale (C-Scale) to measure nurses' confidence in their practice. Responses will be recorded on a five-point Likert scale, ranging from 1 to 5, with 5 indicating "higher confidence." Total scores ranged from 5 to 25, with higher scores indicating greater confidence.

SECONDARY OUTCOMES:
Learning satisfaction | Immediately after intervention.
  This study will use the Indonesian version of the five-item Satisfaction in Learning questionnaire to assess nurses' satisfaction with the assigned learning methods. Responses will be recorded on a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Higher score indicated more satisfied with learning methods.

CONTACTS AND LOCATIONS:
Overall Officials: Nuzul S Hertanti, RN, MS, Principal Investigator — Taipei Medical University
Locations (1):
- Primary Healthcare, Yogyakarta, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No